CLINICAL TRIAL: NCT05518812
Title: Carboprost Tromethamine (Hemabate) for Resection of Fibroids-a Pilot Study
Brief Title: Carboprost (Hemabate) for Fibroid Resection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Chief of Minimally Invasive Gynecologic Surgery in the Department of Obstetrics and Gynecology Albert B. Gerbie, MD, Professor of Obstetrics and Gynecology Professor of Obstetrics and Gynecology (Minimally Invasive Gynecologic Surgery), Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00216433
Record Dates: First submitted 2022-08-05; First posted 2022-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fibroid Uterus; Gynecologic Disease; Leiomyoma, Uterine
MeSH Terms: conditions — Leiomyoma; Genital Diseases, Female | interventions — carboprost tromethamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hemabate (Experimental): Dilute the 250mcg/mL vial with 25mL saline to create a solution of 10mcg/mL, and inject no more than 10mL of diluted solution at the base of the fibroid. The route of administration depends on the location of the fibroid.
  Interventions: Drug: Carboprost Tromethamine

INTERVENTIONS:
Drug: Carboprost Tromethamine — During myomectomy, low-dose carboprost will be injected at the base of the fibroid and repeated as necessary. The efficacy of low-dose carboprost is being assessed, and the total dose administered will not exceed single vial for other indications.
  Other Names: Hemabate

SUMMARY:
The purpose of this research study is to determine if low-dose (i.e., a fraction of what is commonly used) carboprost (Hemabate) helps facilitate fibroid removal (myomectomy).

DETAILED DESCRIPTION:
Uterine fibroids, also known as leiomyomas, are estimated to affect over 80% of women by the time menopause begins. Many women are asymptomatic and remain undiagnosed, therefore the prevalence of the disease is likely underestimated. Leiomyomas are the most common neoplasms to affect women and can cause morbidities such as heavy menstrual bleeding (HMB) and infertility. According to the American College of Obstetricians and Gynecologists, one-fourth of the women with leiomyomas befit treatment, presenting with heavy or prolonged menstrual bleeding, abdominal protrusion, bowel or bladder dysfunction, infertility, recurrent pregnancy loss, painful menses, or pelvic pain. Risk factors associated with developing leiomyomas include: early menarche, use of oral hormonal contraceptives before the age of 16 years, African descent, and an increased body mass index (BMI) (StatPearls Leiomyoma). Factors that may lower the incidence of leiomyomas include: increased parity, use of depot medroxyprogesterone acetate (DMPA) or oral hormonal contraceptives for any duration.

Leiomyomas are benign tumors which arise from monoclonal smooth muscle cells of the uterus (StatPearls Leiomyoma); cells mostly composed of extracellular matrix and encapsulated in a pseudocapsule of areolar tissue. These tumor cells characteristically express higher levels of estrogen and progesterone receptors than normal myometrial cells, and ovarian steroids such as estradiol and progesterone enhance leiomyoma growth. Studies have shown that the size of leiomyomas decrease after menopause when ovarian steroid hormones decline. Leiomyoma cells typically exhibit a low mitotic index. Uterine leiomyomas can impact fertility in multiple ways, for instance, leiomyomas can impede sperm migration, interrupt ovum transport or embryo implantation, and can cause early pregnancy loss. Current treatment options for management of leiomyomas including medical therapies and surgical intervention.

Surgically resecting fibroids is one of the most common procedures performed for women of reproductive age. The goal of surgery is to mitigate symptoms and lower the risk of recurrence. Fibroids identified as FIGO 0 or 1 are typically resected completely at hysteroscopy. Unfortunately, fibroids categorized as FIGO 2 when approached hysteroscopically are almost never completely removed given that there can remain residual leiomyoma within the myometrium that is inaccessible. This commonly requires follow up procedures in the coming 6 months as the myometrial portion migrates into the cavity allowing it to be accessible hysteroscopically. Similarly at laparoscopy/laparotomy, FIGO 6 or 7 fibroids are easily resected completely without significant myometrial disruption. In contrast, FIGO 3-5 fibroids require a much more invasive approach into the myometrium, potentially increasing the risk of uterine rupture during pregnancy, a potentially life-threatening event. Techniques have been developed to promote intraoperative fibroid migration towards the access point (laparoscopy/laparotomy/hysteroscopy) with some success. This is a pilot study to determine whether intramural carboprost at low concentrations can facilitate fibroid migration and minimize the risk of carboprost-related side effects. Using carboprost intraoperatively is relatively simple, does not require additional instrumentation, and potentially results in a more complete resection, reducing operative times and re-operation. With the use of carboprost, the myoma is expelled due to the myometrial contraction, and the leiomyoma is shaved down to the myometrium surface, nullifying the need to deeply invade the myometrium.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo myomectomy with a surgeon in the division of Minimally Invasive Gynecologic Surgery
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* If any oxytocic agents have been or will be administered prior to surgery
* History of renal and/or hepatic impairment
* Active cardiac disease, pulmonary disease, or pelvic inflammatory disease (PID)
* Anemia (Hgb < 7g/dL), diabetes mellitus, jaundice, or epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Does instillation of low-dose carboprost facilitate complete resection of FIGO II fibroids during hysteroscopic resection? | Pre-operatively to 1 month post-operatively
  Pre-operative and post-operative ultrasound will be compared to measure the residual fibroid after hysteroscopic resection with carboprost installation.

SECONDARY OUTCOMES:
To quantitatively assess the efficiency of fibroid resection after carboprost administration by analyzing the video recording from surgery | Through study completion, up to 2 years
  Recordings of all gynecologic surgeries on the site are recorded. The study team members will download and de-identify recordings by removing any PHI and labeling the video with the study ID assigned to the patient by the study team. The video will be used to assess the efficiency of fibroid removal facilitated by low-dose carboprost. The amount of tissue and the time resected will be measured to determine the grams per minute compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy p Milad, MD, MS, Principal Investigator — Northwestern University, Northwestern Memorial Hopsital
Locations (1):
- Northwestern University - Northwestern Medicine, Lavin Family Pavilion, Chicago, Illinois, United States